CLINICAL TRIAL: NCT01706055
Title: Assessment of Strategies for the Management of Flu-like Symptoms in MS Patients Commencing Treatment With Betaferon®
Brief Title: Assessment of Strategies for the Management of Flu-like Symptoms in MS Patients Commencing Treatment With Betaferon (INFLUENCE)
Acronym: INFLUENCE
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 16400; BF1213PL (Other: company internal)
Record Dates: First submitted 2012-09-07; First posted 2012-10-15 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis (MS); Interferon
MeSH Terms: conditions — Multiple Sclerosis | interventions — Interferon beta-1b

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Biological: Interferon beta-1b (Betaseron, BAY86-5046)

INTERVENTIONS:
Biological: Interferon beta-1b (Betaseron, BAY86-5046) — Subcutaneous injections of Betaferon 250 mcg every other day according to Product Characteristic.

SUMMARY:
This will be prospective, multicentre, observational study. Patients who will initiate treatment with IFNβ-1b (Betaferon) will be followed up to 6 months. Baseline visit (visit 0) i.e. treatment initiation plus four follow-up visits (visits 1-4). For each patient demographics, medical history data, safety parameters, presence of flu-like symptoms and measures to prevent or treat these symptoms will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of relapsing-remitting multiple sclerosis (RRMS) according to McDonald (2005) criteria
* Age >/= 18 years old
* Treatment MS patients in whom the attending physician has decided to initiate therapy with interferon beta-1b; Betaferon
* Minimum 6 months wash-out period from previous IFNβ
* Written Informed Consent signed

Exclusion Criteria:

* Patients previously treated with any of the disease modifying drugs (DMDs), with the exception of IFNβ therapy which ended at least 6 months earlier
* Patients receiving treatment with IFN beta other than Betaferon (Bayer)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult MS patients starting Betaferon therapy
Sampling Method: Non-Probability Sample
Enrollment: 629 (Actual)
Dates: Start 2012-09; Primary Completion 2015-09 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Mean severity score of Flu-Like Symptoms (FLS) recorded within the first 6 months following treatment initiation | 6 months
MS patient with Flu-Like Symptoms (FLS) demographic profile | Up to 1 month
  For demographic assessment the following parameters will be recorded at visit 0: birthdate (at least year), sex, weight, height.
Frequency of usage of particular pharmacological and non-pharmacological practices applied by investigators to prevent or manage FLS | 6 months

SECONDARY OUTCOMES:
The impact of FLS on patients daily activities as measured by current professional/educational status | From baseline up to 6 months
Betaferon tolerability measured as occurrence of Adverse Events (AE) and FLS over 6 months period | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Poland